CLINICAL TRIAL: NCT00199316
Title: Postoperative Pain Control After Kidney Surgery : a Comparison of Intrathecal Morphine Plus PCA and PCA Only
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I48015
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2007-10

CONDITIONS: Postoperative Pain
Keywords: patient who recieve kidney surgery and Patient controlled anesthesia with spinal morphine, intrathecal
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: spinal morphine

SUMMARY:
postoperative pain after kidney surgery is very high. We always use PCA for postopertive pain. But almost patients still had severe pain. We try to use spinal morphine before operation aims to reduce pain.

ELIGIBILITY:
Inclusion Criteria:

* kidney surgery who less than 60 years old.
* no underlying disease
* ASA less than 3

Exclusion Criteria:

* refuse spinal morphine
* history of morphine allery

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-01; Study Completion 2005-11

PRIMARY OUTCOMES:
pain score | 48 hours

SECONDARY OUTCOMES:
morphine consumption in PCA | 48 hours
side effect | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Polpun Boonmak, MD, Study Director — lecturer in Khon Kaen University
Locations (1):
- Khon Kaen university, Srinagarind Hospital, Muang, Changwat Khon Kaen, Thailand